CLINICAL TRIAL: NCT05166434
Title: Radiographic Assessment of Crestal Maxillary Sinus Membrane Elevation Using Different Dental Implant Heights in Atrophic Posterior Maxilla
Brief Title: Assessment Crestal Maxillary Sinus Membrane Elevation Using Different Implant Heights
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maher Mohammed Hebah Maqbol, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: o m f s 335
Record Dates: First submitted 2021-12-07; First posted 2021-12-22 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Bone Formation Around Implant After Crestal Sinus Lifting
Keywords: Stability, implant. sinus lifting, bone formation

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- bone formation around implant at 2mm membrane elevation crestal sinus lifting (Active Comparator)
  Interventions: Procedure: trans-crestal sinus lifting
- bone formation around implant at 4mm membrane elevation crestal sinus lifting (Active Comparator)
  Interventions: Procedure: trans-crestal sinus lifting
- bone formation around implant at 6mm membrane elevation crestal sinus lifting (Active Comparator)
  Interventions: Procedure: trans-crestal sinus lifting

INTERVENTIONS:
Procedure: trans-crestal sinus lifting — this study will be divided in to three different groups, each group will receive a same technique of Crestal maxillary sinus lifting and implant placement at 2,4,6 mm heights.
  Other Names: Closed sinus lifting

SUMMARY:
This study is aiming to evaluate primary stability and bone gain in trans-crestal osseodencification technique using Regular concaved osteotomes at different height elevations.

DETAILED DESCRIPTION:
For those patient who need up to 2-6 mm of vertical height, the 1-stage transcrestal osteotome technique shown to be stable over long term.

The most important negative factor that can be inferred from the results is that BAOSFE becomes less predictable when there is 4 mm or less of preexisting alveolar bone height beneath the sinus. Moreover, more challenging situation is the magnitude of tapping force, which may accidently perforate the antral membrane causing a lot of complication in the naso-antral apparatus by excessive taping force. The expansion of the osteotomy sites is performed with a number of Concave tipped tapered osteotomes with increasing diameters that are applied through the edentulous alveolar crest at the inferior border of the maxillary sinus floor. With each insertion of a larger osteotome, bone is compressed, pushed laterally and apically while pushing the garnered bone apically beneath the tented membrane.

ELIGIBILITY:
Inclusion Criteria:

* Patients with edentulous vertically deficient posterior maxillary ridge a minimum 4 mm height of alveolar bone, and 6 mm in width.
* Both males as well as females without any active periodontal disease.
* All patients are in a good health with no systemic, immunologic or debilitating diseases that could affect normal bone healing.
* All selected patients are non-smokers and non-alcoholics.
* Patients are free from T.M.J troubles, abnormal oral habits such as bruxism.
* The edentulous ridges are covered with optimal thickness of mucoperiosteum with no signs of inflammation, ulceration or scar tissue.
* Remaining natural teeth have good periodontal tissue support and occlusion showed sufficient inter arch space for future prosthesis.

Exclusion Criteria:

1. On the local level, patients with maxillary sinus diseases, former sinus surgery and unfavorable inter maxillary relationship will be excluded.
2. General contraindications to implant surgery.
3. Subjected to irradiation in the head and neck area less than 1 year before implantation.
4. Untreated periodontitis.
5. Poor oral hygiene and motivation.
6. Uncontrolled diabetes.
7. Pregnant or nursing.
8. Substance abuse.
9. Psychiatric problems or unrealistic expectations.
10. Severe bruxism or clenching.
11. Immunosuppressed or immunocompromised.
12. Treated or under treatment with intravenous amino-bisphosphonates.
13. Lack of opposite occluding dentition/prosthesis in the area intended for implant placement.
14. Active infection or severe inflammation in the area intended for implant placement.
15. Need of bone augmentation procedures at implant placement.
16. Unable to open mouth sufficiently to accommodate the surgical tooling.
17. Patients participating in other studies, if the present protocol could not be properly followed.
18. Referred only for implant placement or unable to attend a 5-year follow-up.
19. Requiring only single implant-supported crowns.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Measuring bone formation and density beyond apical part of dental implant after closed sinus lifting | 4 months after Dental implant placement
  CBCT superimposition of the Pre-operative and Post-operative

SECONDARY OUTCOMES:
Measuring secondary stability of dental implants | 4 months after Dental implant placement
  osttell device (ISQ)

CONTACTS AND LOCATIONS:
Locations (1):
- Maher Mohammed Hebah Maqbol, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No